CLINICAL TRIAL: NCT02140333
Title: Phase 3 Study of Erlotinib 100mg or 150mg in Treating EGFR Mutated Patients With Non-small Cell Lung Cancer
Brief Title: Erlotinib 100mg or 150mg in Treating EGFR Mutated NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, The First Affiliated Hospital of Guangzhou Medical Univers, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAHG20130819; GZMC201301
Record Dates: First submitted 2013-10-05; First posted 2014-05-16 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: NSCLC; EGFR Mutation
Keywords: erlotinib; EGFR mutation
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib 100mg (Experimental): Erlotinib 100mg
  Interventions: Drug: Erlotinib
- Erlotinib 150mg (Active Comparator): Erlotinib 150mg
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — 100mg vs. 150mg
  Other Names: tarceva

SUMMARY:
The purpose of this study is to determine whether 100mg erlotinib had similar effect compared with 150mg erlotinib in NSCLC patients with EGFR mutation in China.

DETAILED DESCRIPTION:
In China it was confirmed that 150mg Erlotinib was effective in NSCLC patients wtih EGFR mutation, but reducing dose occurring in some patients because of the drug related side-effects. Thus, we sought to investigate that in Chinese patients with EGFR mutation whether low dose (100mg) Erlotinib had similar efficacy but lower toxcities compared with standad dose (150mg) Erlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of NSCLC with phase IIIB or IV disease;
2. Sensitive mutation EGFR gene (18, 19 del, 21 L858R gene mutation) (mutation detection methods:ARMS-PCR, sequence method)
3. Never received anti-tumor therapies for the advanced stage;
4. Never used EGFR inhibitors;
5. Measurable disease by RECIST criteria;
6. Male or female patients >=18 years of age;
7. ECOG karnofsky performance 0~3, life expectancy is greater than 12 weeks;
8. Patients must be accessible for treatment and follow-up;

Exclusion Criteria:

1. Previously used EGFR inhibitors
2. Mix ingredients in patients with squamous cell carcinoma, small cell lung cancer;
3. Allergic to erlotinib;
4. Non-measurable lesions
5. Pregnant or lactating women;
6. Patients having other factors that preventing researchers from enrollment them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years after the initial dose

SECONDARY OUTCOMES:
The objective response rate | Patients will be followed for an expected average of 6 months

OTHER OUTCOMES:
Overall survival | 3 year after the initial dose
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou medical university, Guanzhou, Guangdong, China